CLINICAL TRIAL: NCT00859534
Title: A Phase II, Open Label Pilot Study to Evaluate the Safety and Efficacy of A Bioresorbable Subcutaneous Implant of CUV1647 in Patients With Solar Urticaria (SU)
Brief Title: Phase II Solar Urticaria (SU) Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clinuvel Pharmaceuticals Limited (Industry)
Responsible Party: Dr Dennis Wright, Clinuvel Pharmaceuticals Limitied
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CUV016
Record Dates: First submitted 2009-03-05; First posted 2009-03-11 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Solar Urticaria
Keywords: Solar Urticaria
MeSH Terms: conditions — Urticaria, Solar | interventions — afamelanotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: afamelanotide — 16mg afamelanotide, one dose for the duration of the clincial trial

SUMMARY:
Urticaria is one of the most common dermatological conditions with diverse clinical presentations and causes. Solar urticaria (SU) is a rare subset of physical urticaria, where symptoms are induced by direct exposure of the skin to sunlight. As little as 5 minutes of sun exposure can cause flares and whealing on exposed skin sites, accompanied by severe itching. The wavelengths of radiation causing the eruption (i.e. the action spectrum) are in the ultraviolet or visible light range. Initially described by Merklen in 1904, SU may have a very sudden and dramatic onset, and then rapidly disappear once the exposure ceases. A delayed form of SU has also been reported, although this is extremely rare. Information on the pathophysiology of SU is limited and symptoms are confined to areas of the body exposed to direct sunlight. The condition can be very distressing and severely impair the individual's ability to go outdoors and to tolerate indoor lighting. The standard therapy, i.e. oral antihistamines, is only partially effective and may provide little worthwhile relief of symptoms.

This pilot study is proposed to evaluate implants containing 16mg CUV1647 as a prophylactic treatment for patients with SU. The effectiveness of CUV1647 will be assessed by determining the minimum urticarial dose before and after treatment.

DETAILED DESCRIPTION:
When human skin is exposed to ultraviolet radiation from the sun or via the use of solaria, it responds by increasing melanin levels within epidermal melanocytes. Ultraviolet light enhances the local production and release of alpha-melanocyte stimulating hormone (alpha-MSH), which results in increased melanin levels through a process known as melanogenesis. Melanin, in the form of eumelanin, is a photoprotective agent. The mechanisms proposed for photoprotection include, but are not limited to, the absorption and scattering of UV and visible radiation, free radical scavenging and quenching of UV light. There is also increasing evidence that melanogenesis represents a major antioxidant defence mechanism in melanocytes, neutralising the deleterious effects of free radicals and active oxygen species. Eumelanin acts as a neutral density filter and, unlike most sunscreens, reduces all wavelengths of light equally so that the photoprotection provided by epidermal melanin pigmentation is essentially independent of wavelength.

CUV1647 ([Nle4-D-Phe7]-alpha-MSH) is a potent and longer lasting analogue of alpha-MSH which stimulates the production of eumelanin in the skin without the specific cell damage that usually occurs when melanin production is stimulated by UV radiation.

Urticaria is one of the most common dermatological conditions with diverse clinical presentations and causes. Solar urticaria (SU) is a rare subset of physical urticaria, where symptoms are induced by direct exposure of the skin to sunlight. As little as 5 minutes of sun exposure can cause flares and whealing on exposed skin sites, accompanied by severe itching. The wavelengths of radiation causing the eruption (i.e. the action spectrum) are in the ultraviolet or visible light range. Initially described by Merklen in 1904, SU may have a very sudden and dramatic onset, and then rapidly disappear once the exposure ceases. A delayed form of SU has also been reported, although this is extremely rare. Information on the pathophysiology of SU is limited and symptoms are confined to areas of the body exposed to direct sunlight. The condition can be very distressing and severely impair the individual's ability to go outdoors and to tolerate indoor lighting. The standard therapy, i.e. oral antihistamines, is only partially effective and may provide little worthwhile relief of symptoms.

This pilot study is proposed to evaluate implants containing 16mg CUV1647 as a prophylactic treatment for patients with SU. The effectiveness of CUV1647 will be assessed by determining the minimum urticarial dose before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with a diagnosis of solar urticaria (confirmed by phototesting) of sufficient severity that they have requested treatment to alleviate symptoms.
* React to provocation with a light source
* Aged 18-70 years
* Fitzpatrick Skin Type I- IV
* Written informed consent prior to the performance of any study-specific procedure.

Exclusion Criteria:

* Allergy to CUV1647 or the polymer contained in the implant
* Any co-existent photodermatosis such as polymorphic light eruption (PLE), discoid lupus erythematosus (DLE) or erythropoietic porphyria (EPP).
* Personal history of melanoma, lentigo maligna or multiple (3 or more) dysplastic nevi.
* Current Bowen's disease, basal cell carcinoma, squamous cell carcinoma, or other malignant or premalignant skin lesions.
* Diagnosed with HIV/AIDS or hepatitis.
* Any evidence of organ dysfunction or deviation from normal the clinical or laboratory determinations judged to be clinically significant by the Investigator.
* History of disorders of the gastrointestinal, hepatic, renal, cardiovascular, respiratory, endocrine (including diabetes, Cushing's syndrome, Addison's disease, Peutz-Jeagher syndrome), neurological (including seizures), haematological (especially anaemia of less than 10 g/100 mL) or systemic disease judged to be clinically significant by the Investigator.
* Acute history of drug or alcohol abuse (in the last 12 months).
* Major medical or psychiatric illness.
* Patient assessed as not suitable for the study in the opinion of the investigator (e.g. noncompliance history, allergic to local anaesthetics, faints when given injections or giving blood).
* Female who is pregnant (confirmed by positive serum β-HCG pregnancy test prior to baseline) or lactating.
* Females of child-bearing potential (pre-menopausal, not surgically sterile) not using adequate contraceptive measures (i.e. oral contraceptives, diaphragm plus spermicide, intrauterine device).
* Sexually active men with partners of child bearing potential not using barrier contraception during the trial and for a period of three months hereafter.
* Participation in a clinical trial for an investigational agent within 30 days prior to the screening visit.
* Any factors that may affect skin reflectance measurements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-12; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To determine whether a CUV1647 (synthetic alpha-MSH analogue) bioresorbable implant can reduce the susceptibility of patients with Solar Urticaria to provocation with a standardized light source (measured as a change in minimum urticarial dose, (MUD)). | 60 days

SECONDARY OUTCOMES:
To evaluate the safety/tolerability of CUV1647 by measuring treatment-emergent adverse events. | 60 days
To determine the effect of CUV1647 on melanin density at several specified body sites. | 60 days
To evaluate a change in the MUD between Days 30 and 60. | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Lesley Rhodes, M.D., Principal Investigator — Salford Royal Foundation Hospital (Hope Hospital)
Locations (1):
- Salford Royal Foundation Hospital (Hope Hospital), Manchester, United Kingdom